CLINICAL TRIAL: NCT07311902
Title: Comparison of Patient Satisfaction Survey and Pain Follow-up in Patients Who Underwent M-Tapa Block and Transversus Abdominal Plane Block for Postoperative Analgesia in Unilateral Open Inguinal Hernia Repair Surgery
Brief Title: M-Tapa Block and Transversus Abdominal Plane Block for Postoperative Analgesia in Unilateral Open Inguinal Hernia Repair Surgery
Acronym: pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Omer Doymus, assistant professor, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B.30.2.YYU.0.01.00.00/93
Record Dates: First submitted 2025-06-18; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-06

CONDITIONS: Pain Management; Mtapa Block; TAP Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Active Comparator): The block needle will be advanced to the fascial plane between the internal oblique and transversus abdominis muscles by placing the USG transversely on the mid-axillary line between the iliac crest and subcostal planes. 5 ml saline will be injected and the block location will be confirmed. After the block location is confirmed, a total of 20 ml of 0.25% bupivacaine will be injected unilaterally and the procedure will be completed.
  Interventions: Procedure: TAP Block Group
- Group M (Active Comparator): Using the in-plane technique, the probe will be pushed slightly to visualize the lower part of the costochondral angle at the central level, the block needle will be advanced in the caudal-cranio direction, 5 ml of saline will be injected into the layer between the transverse abdominal muscle and the lower plane of the costal cartilage via a 22G 100 mm block needle and the block location will be confirmed. After the block location is confirmed, a total of 20 ml of 0.25% bupivacaine will be injected unilaterally and the procedure will be completed.
  Interventions: Procedure: M TAPA block

INTERVENTIONS:
Procedure: TAP Block Group — 20 ml of 0.25% bupivacaine
  Arms: Group T
Procedure: M TAPA block — 20 ml of 0.25% bupivacaine
  Arms: Group M

SUMMARY:
Patients will be called to the operating room one hour before surgery and no premedication will be applied before coming to the operating room. Patients in both groups who are taken to the block room will be administered 1-2 mg iv midazolam for sedation. M TAPA block will be applied for the surgical procedure. After aseptic conditions are provided, the high-frequency linear US probe will be covered with a sterile sheath. The US probe will be placed in the saggital plane at the costochondral angle where the midclavicular line intersects the costal cartilage. 5 ml of saline will be injected using the in-plane technique using a 22G 100 mm block needle and the block location will be verified. After the block location is verified, a total of 20 ml of 0.25% bupivacaine will be injected unilaterally and the procedure will be terminated. After aseptic conditions are provided, the high-frequency linear US probe will be covered with a sterile sheath. In TAP block, the block needle will be advanced to the fascial plane between the internal oblique and transversus abdominis muscles with the in-plane technique and the procedure will be completed by injecting 5 ml 20 ml 0.25% bupivacaine unilaterally. The same analgesia protocol will be applied to both groups intraoperatively and postoperatively, and a survey will be conducted on the patients at the 24th hour postoperatively.

ELIGIBILITY:
Exclusion Criteria:

* History of bleeding diathesis
* Allergy or sensitivity to local anesthetics and opioids
* Infection in the area where the block will be applied
* Alcohol or drug addiction
* Patients with a BMI > 30
* Suspected pregnancy
* Women in pregnancy or lactation
* Patients with allergies to study drugs
* Patient refusal
* Use of anticoagulant agents

Inclusion Criteria:

* Planning for elective unilateral open inguinal hernia repair surgery
* ASA I-II status
* Being between 18 and 65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
pain score | The primary aim of our study was to compare VAS scores at 1, 2, 4, 8, 12, and 24 hours postoperatively and to evaluate the level of comfort.
  Patients' pain scores will be evaluated

SECONDARY OUTCOMES:
The QoR-15 Patient Questionnaire, a 40-question global recovery rating system with a Turkish variant | 24 hours following surgery.
  To compare patient satisfaction survey and pain monitoring in patients who underwent M-Tapa Block and Transversus Abdominal Plane block for postoperative analgesia in unilateral open inguinal hernia repair surgery and to suggest a more effective method.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Regional Education and Research Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No